CLINICAL TRIAL: NCT01795547
Title: A 28-week, Randomised, Open-label Study Evaluating the Effectiveness of Aripiprazole Once-monthly Versus Paliperidone Palmitate in Adult Patients With Schizophrenia
Brief Title: Aripiprazole Once-monthly Versus Paliperidone Palmitate in Adult Patients With Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Collaborators: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14724A; 2012-002785-12 (EudraCT Number)
Record Dates: First submitted 2013-02-18; First posted 2013-02-20 (Estimated); Results first posted 2015-12-03 (Estimated); Last update posted 2017-03-17 (Actual); Status verified 2017-02

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Aripiprazole; Paliperidone Palmitate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aripiprazole and aripiprazole once-monthly (Experimental)
  Interventions: Drug: Aripiprazole and aripiprazole once-monthly
- Paliperidone and paliperidone palmitate (Active Comparator)
  Interventions: Drug: Paliperidone and paliperidone palmitate

INTERVENTIONS:
Drug: Aripiprazole and aripiprazole once-monthly — Oral aripiprazole tablets according to Summary of Product Characteristics (SmPC)/United States Prescription Information (USPI) daily for 4 weeks followed by the 1st aripiprazole intramuscular (IM) injection at the end of Week 4. Oral tablets were taken for 2 more weeks after the 1st injection. Starting at the end of Week 8, additional injections were given every 4 weeks until Week 24.
  Other Names: Aripiprazole: Abilify®; Aripiprazole (extended-release injectable suspension): Abilify Maintena®
  Arms: Aripiprazole and aripiprazole once-monthly
Drug: Paliperidone and paliperidone palmitate — Oral paliperidone tablets according to SmPC/USPI daily for 3 weeks followed by 2 paliperidone palmitate IM injections at Weeks 3 and 4, respectively. Starting at the end of Week 8, additional injections were given every 4 weeks until Week 24.
  Other Names: Paliperidone: Invega®; Paliperidone palmitate: Xeplion® or Invega® Sustenna®
  Arms: Paliperidone and paliperidone palmitate

SUMMARY:
To assess the effectiveness of aripiprazole once-monthly in the maintenance treatment of patients with a diagnosis of schizophrenia as defined by the Diagnostic and Statistical Manual of Mental Disorders, 4th edition, Text Revision (DSM-IV-TR®), in a naturalistic care setting by comparing it to an existing long-acting antipsychotic, paliperidone palmitate.

ELIGIBILITY:
Main Inclusion Criteria:

* The patient has schizophrenia, diagnosed according to DSM-IV-TR®.
* The patient has a CGI-S score from mildly ill to markedly ill at the Screening and Baseline Visit(s).
* The patient is in need of a change in the current antipsychotic treatment and in the judgement of the investigator the patient would benefit from an extended treatment with a once-monthly formulation.
* The patient agrees to protocol-defined use of effective contraception.

Main Exclusion Criteria:

* The patient has any current psychiatric disorder or Axis I disorder (DSM-IV® criteria) other than schizophrenia established as the primary diagnosis.
* The patient is experiencing acute exacerbation of psychotic symptoms at the Screening Visit or between the Screening and Baseline Visits.
* The patient in the investigator's judgment has shown significant intolerance and/or lack of efficacy to oral aripiprazole, paliperidone or risperidone.
* The patient is at significant risk of harming himself/herself or others according to the investigator's judgement or according to Columbia-Suicide Severity Rating Scale (C-SSRS).
* The patient has a history of neuroleptic malignant syndrome.
* The patient has or has had significant medical condition that would expose him or her to an undue risk of a significant adverse event or interfere with assessments of safety or efficacy during the course of the study including, but not limited to neurological, hepatic, renal, metabolic, haematological, immunological, gastrointestinal, pulmonary, or cardiovascular disorders.
* The patient has a disease or takes medication that could, in the investigator's opinion, interfere with the assessments of safety, tolerability, or efficacy, or interfere with the conduct or interpretation of the study.
* The patient is, in the investigator's opinion, unlikely to comply with the protocol or is unsuitable for any reason.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 295 (Actual)
Dates: Start 2013-02; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com
Locations (2):
- United States (2):
  - US002, Los Angeles, California
  - US006, San Diego, California

REFERENCES:
- [Derived] Potkin SG, Loze JY, Forray C, Baker RA, Sapin C, Peters-Strickland T, Beillat M, Nylander AG, Hertel P, Nitschky Schmidt S, Eramo A, Hansen K, Naber D. Multidimensional Assessment of Functional Outcomes in Schizophrenia: Results From QUALIFY, a Head-to-Head Trial of Aripiprazole Once-Monthly and Paliperidone Palmitate. Int J Neuropsychopharmacol. 2017 Jan 1;20(1):40-49. doi: 10.1093/ijnp/pyw093. PMID 27927736
- [Derived] Naber D, Hansen K, Forray C, Baker RA, Sapin C, Beillat M, Peters-Strickland T, Nylander AG, Hertel P, Andersen HS, Eramo A, Loze JY, Potkin SG. Qualify: a randomized head-to-head study of aripiprazole once-monthly and paliperidone palmitate in the treatment of schizophrenia. Schizophr Res. 2015 Oct;168(1-2):498-504. doi: 10.1016/j.schres.2015.07.007. Epub 2015 Jul 29. PMID 26232241
- See also: EMA EudraCT Results: 2012-002785-12 — https://www.clinicaltrialsregister.eu/ctr-search/trial/2012-002785-12/results

RESULTS

PARTICIPANT FLOW:
Groups:
- Aripiprazole: Aripiprazole and aripiprazole once-monthly: Oral aripiprazole tablets according to Summary of Product Characteristics (SmPC)/United States Prescription Information (USPI) daily for 4 weeks followed by the 1st aripiprazole intramuscular (IM) injection. Oral tablets will be taken for 2 more weeks after the 1st injection. Additional injections every 4 weeks until Week 24
- Paliperidone: Paliperidone and paliperidone palmitate: Oral paliperidone tablets according to SmPC/USPI daily for 3 weeks followed by paliperidone palmitate IM injections every 4 weeks with last dose at Week 24 according to SmPC/USPI
Period: Overall Study
Arm/Group | Aripiprazole | Paliperidone
Started | 148 | 147
Completed | 100 | 83
Not Completed | 48 | 64
Not completed — Adverse Event | 16 | 27
Not completed — Lack of Efficacy | 8 | 3
Not completed — Protocol Violation | 6 | 4
Not completed — Lost to Follow-up | 2 | 5
Not completed — Withdrawal of consent | 7 | 12
Not completed — Not Treated | 4 | 10
Not completed — Non-compliance with IMP | 1 | 1
Not completed — Others | 4 | 1
Not completed — Not stated | 0 | 1

BASELINE CHARACTERISTICS:
Population: Demographic data is based on all enrolled subjects, which were also all randomized
Groups:
- Total: Total of all reporting groups
Arm/Group | Aripiprazole | Paliperidone | Total
Number analyzed (Participants) | 148 | 147 | 295
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.6 (10.83) | 41.0 (10.87) | 41.8 (10.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 59 | 118
  Male | 89 | 88 | 177
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 44 | 38 | 82
  White | 102 | 102 | 204
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 4 | 5

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 28 in Quality of Life Scale (QLS) Total Score
Description: The QLS is a clinician-rated scale designed to assess deficit symptoms of schizophrenia and functioning during the preceding 4 weeks. The QLS consists of 21 items in 4 domains: Interpersonal Relations (eight items), Instrumental Role (four items), Intrapsychic Foundations (seven items), and Common Objects and Activities (two items). Each item was rated on a 7-point scale, from 0 (severe impairment) to 6 (normal or unimpaired functioning). Definitions were provided for 4 anchor points of the 7 points. Each item had a brief description of the judgement to be made and a set of suggested probes for the clinician. The total score was calculated as the sum of all 21 items giving a range of 0 to 126, where the higher score indicated normal or unimpaired functioning.
Time Frame: Baseline, Week 28
Population: Effectiveness data is based on all patients who received study medicine, who had a valid baseline assessment, and at least 1 valid post-baseline assessment of the QLS (Full analysis set). Effectiveness was measured at Weeks 0, 4, 8, 16, and 28.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Aripiprazole: Oral aripiprazole tablets according to Summary of Product Characteristics (SmPC)/United States Prescription Information (USPI) daily for 4 weeks followed by the 1st aripiprazole intramuscular (IM) injection at the end of Week 4. Oral tablets were taken for 2 more weeks after the 1st injection. Starting at the end of Week 8, additional injections were given every 4 weeks until Week 24.
- Paliperidone: Oral paliperidone tablets according to SmPC/USPI daily for 3 weeks followed by 2 paliperidone palmitate IM injections at Weeks 3 and 4, respectively. Starting at the end of Week 8, additional injections were given every 4 weeks until Week 24.
Arm/Group | Aripiprazole | Paliperidone
Number analyzed (Participants) | 136 | 132
units on a scale | 7.47 (1.53) | 2.80 (1.62)
Statistical Analysis 1: Comparison: Aripiprazole vs Paliperidone; Comparison of aripiprazole versus paliperidone was made using estimates from a mixed model for repeated measurements (MMRM) using an unstructured covariance matrix; Test type: Non-Inferiority or Equivalence — Non-inferiority of the primary endpoint was considered confirmed if the lower bound of the 2-sided 95% CI at Week 28 was > -5 or equivalently if the p-value for the 1-sided test of H0: D ≤ -5 against H1: D > -5 was ≤2.5%, where D was the mean treatment difference (aripiprazole minus paliperidone). Superiority was then tested as pre-specified with the FAS and demonstrated for aripiprazole over paliperidone, since the lower bound of the 95% CI was >0; p = 0.036, Mixed Models Analysis; The model uses an unstructured variance/covariance matrix; Least Squares Mean Difference = 4.666, 95% CI 2-sided [0.316 to 9.015]

2. Secondary Outcome: Investigator's Assessment Questionnaire (IAQ) Total Score at Week 28
Description: The IAQ is a clinician-rated scale designed to assess the relative effectiveness (efficacy, safety and tolerability) of antipsychotic medications in patients with schizophrenia or schizoaffective disorder. The IAQ consists of 12 items: positive symptoms, negative symptoms, other efficacy symptoms, cognition, energy, mood, somnolence, weight gain, signs and symptoms of prolactin elevation, akathisia, EPS (other than akathisia) and other safety or tolerability issues. For each item, the current medication was compared with previous antipsychotic medication on a five-point scale from 1 (Much better) to 5 (Much worse), or that item is Not applicable. The sum of the 12 items ranged from 12 (the current medication was much better than previous antipsychotic medication) to 60 (the current medication was much worse than previous antipsychotic medication).
Time Frame: Week 28
Population: Effectiveness data is based on all patients who received study medicine, who had a valid baseline assessment, and at least 1 valid post-baseline assessment of the QLS (Full analysis set). Effectiveness was measured at Weeks 4, 8, 16, and 28. Since the IAQ was assessed from week 4, the analysis was based on 133 and 131 patients
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Aripiprazole | Paliperidone
Number analyzed (Participants) | 133 | 131
units on a scale | 32.32 (0.52) | 33.81 (0.55)
Statistical Analysis 1: Comparison: Aripiprazole vs Paliperidone; Test type: Superiority or Other; p = 0.043, Mixed Models Analysis — All secondary endpoints were tested without any hierarchical testing strategy and no adjustment for multiplicity; The model uses an unstructured variance/covariance matrix; Least Squares Mean Difference = -1.492, 95% CI 2-sided [-2.935 to -0.049]

3. Secondary Outcome: Change From Baseline to Week 28 in CGI-S Score
Description: Clinical Global Impression - Severity of Illness (CGI-S) score provides the clinician's impression of the patient's current state of mental illness. The clinician uses his or her clinical experience of this patient population to rate the severity of the patient's current mental illness on a 7-point scale ranging from 1 (normal - not at all ill) to 7 (among the most extremely ill patients).
Time Frame: Baseline, Week 28
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Aripiprazole | Paliperidone
Number analyzed (Participants) | 136 | 132
units on a scale | -0.75 (0.07) | -0.46 (0.07)
Statistical Analysis 1: Comparison: Aripiprazole vs Paliperidone; Test type: Superiority or Other; p = 0.004, Mixed Models Analysis — All secondary endpoints were tested without any hierarchical testing strategy and no adjustment for multiplicity; The model uses an unstructured variance/covariance matrix; Least Squares Mean Difference = -0.283, 95% CI 2-sided [-0.477 to -0.090]

4. Secondary Outcome: Change From Baseline to Week 28 in the 'Common Objects and Activities' QLS Domain Score
Description: The QLS is a clinician-rated scale designed to assess deficit symptoms of schizophrenia and functioning during the preceding 4 weeks. The QLS consists of 21 items in 4 domains: Interpersonal Relations (eight items), Instrumental Role (four items), Intrapsychic Foundations (seven items), and Common Objects and Activities (two items). Each item was rated on a 7-point scale, from 0 (severe impairment) to 6 (normal or unimpaired functioning). The Common Objects and Activities domain score was calculated as the sum of 2 items (numbers 18 and 19) giving a range of 0 to 12, where the higher score indicated less unimpaired functioning.
Time Frame: Baseline, Week 28
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Aripiprazole | Paliperidone
Number analyzed (Participants) | 136 | 132
units on a scale | 0.52 (0.16) | 0.18 (0.17)
Statistical Analysis 1: Comparison: Aripiprazole vs Paliperidone; Test type: Superiority or Other; p = 0.149, Mixed Models Analysis — All secondary endpoints were tested without any hierarchical testing strategy and no adjustment for multiplicity; The model uses an unstructured variance/covariance matrix; Least Squares Mean Difference = 0.331, 95% CI 2-sided [-0.120 to 0.782]

5. Secondary Outcome: Change From Baseline to Week 28 in the 'Intrapsychic Foundations' QLS Domain Score
Description: The QLS is a clinician-rated scale designed to assess deficit symptoms of schizophrenia and functioning during the preceding 4 weeks. The QLS consists of 21 items in 4 domains: Interpersonal Relations (eight items), Instrumental Role (four items), Intrapsychic Foundations (seven items), and Common Objects and Activities (two items). Each item was rated on a 7-point scale, from 0 (severe impairment) to 6 (normal or unimpaired functioning). The Intrapsychic Foundations domain score was calculated as the sum of 7 items (numbers 13 to 17 and 20 and 21) giving a range of 0 to 42, where the higher score indicated less unimpaired functioning.
Time Frame: Baseline, Week 28
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Aripiprazole | Paliperidone
Number analyzed (Participants) | 136 | 132
units on a scale | 2.25 (0.59) | 0.50 (0.63)
Statistical Analysis 1: Comparison: Aripiprazole vs Paliperidone; Test type: Superiority or Other; p = 0.039, Mixed Models Analysis — All secondary endpoints were tested without any hierarchical testing strategy and no adjustment for multiplicity; The model uses an unstructured variance/covariance matrix; Least Squares Mean Difference = 1.753, 95% CI 2-sided [0.093 to 3.412]

6. Secondary Outcome: Change From Baseline to Week 28 in the 'Interpersonal Relations' QLS Domain Score
Description: The QLS is a clinician-rated scale designed to assess deficit symptoms of schizophrenia and functioning during the preceding 4 weeks. The QLS consists of 21 items in 4 domains: Interpersonal Relations (eight items), Instrumental Role (four items), Intrapsychic Foundations (seven items), and Common Objects and Activities (two items). Each item was rated on a 7-point scale, from 0 (severe impairment) to 6 (normal or unimpaired functioning). The Interpersonal Relations domain score was calculated as the sum of 8 items (numbers 1 to 8) giving a range of 0 to 48, where the higher score indicated less unimpaired functioning.
Time Frame: Baseline, Week 28
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Aripiprazole | Paliperidone
Number analyzed (Participants) | 136 | 132
units on a scale | 3.24 (0.68) | 1.47 (0.72)
Statistical Analysis 1: Comparison: Aripiprazole vs Paliperidone; Test type: Superiority or Other; p = 0.070, Mixed Models Analysis — All secondary endpoints were tested without any hierarchical testing strategy and no adjustment for multiplicity; The model uses an unstructured variance/covariance matrix; Least Squares Mean Difference = 1.764, 95% CI 2-sided [-0.143 to 3.672]

7. Secondary Outcome: Change From Baseline to Week 28 in the 'Instrumental Role' QLS Domain Score
Description: The QLS is a clinician-rated scale designed to assess deficit symptoms of schizophrenia and functioning during the preceding 4 weeks. The QLS consists of 21 items in 4 domains: Interpersonal Relations (eight items), Instrumental Role (four items), Intrapsychic Foundations (seven items), and Common Objects and Activities (two items). Each item was rated on a 7-point scale, from 0 (severe impairment) to 6 (normal or unimpaired functioning). The Instrumental Role domain score was calculated as the sum of 4 items (numbers 9 to 12) giving a range of 0 to 24, where the higher score indicated less unimpaired functioning.
Time Frame: Baseline, Week 28
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Aripiprazole | Paliperidone
Number analyzed (Participants) | 136 | 132
units on a scale | 1.76 (0.42) | 0.83 (0.45)
Statistical Analysis 1: Comparison: Aripiprazole vs Paliperidone; Test type: Superiority or Other; p = 0.130, Mixed Models Analysis — All secondary endpoints were tested without any hierarchical testing strategy and no adjustment for multiplicity; The model uses an unstructured variance/covariance matrix; Least Squares Mean Difference = 0.922, 95% CI 2-sided [-0.275 to 2.119]

8. Secondary Outcome: Change From Baseline to Week 28 in SWN-S Total Score
Description: The SWN-S is a patient-rated scale designed to measure subjective effects of neuroleptic drugs to psychopathology, quality of life, and compliance over the past 7 days. The 20 items (10 positive and 10 negative statements) are grouped in 5 subscales (mental functioning, self-control, physical functioning, emotional regulation and social integration). Each subscale contains 4 items. Each item was rated on a six-point Likert scale, from not at all to very much. A score was calculated for each subscale, and the total score ranged from 20 to 120, where the higher score indicated better well-being.
Time Frame: Baseline, Week 28
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Aripiprazole | Paliperidone
Number analyzed (Participants) | 136 | 132
units on a scale | 4.82 (1.24) | 3.81 (1.31)
Statistical Analysis 1: Comparison: Aripiprazole vs Paliperidone; Test type: Superiority or Other; p = 0.561, Mixed Models Analysis — All secondary endpoints were tested without any hierarchical testing strategy and no adjustment for multiplicity; The model uses an unstructured variance/covariance matrix; Least Squares Mean Difference = 1.007, 95% CI 2-sided [-2.402 to 4.417]

9. Secondary Outcome: Change From Baseline to Week 28 in the TooL Total Score
Description: Tolerability and Quality of Life (TooL) is a patient-rated scale developed to measure the impact of side-effects on the quality of life in patients treated with antipsychotic medication. The TooL consists of 8 domains: mood (worry-upset), function capabilities, fatigue-weakness, weight gain, stiffness-tremor, physical restlessness, sexual dysfunction, and dizziness-nausea. Each domain was rated on a four-point scale from 1 (no impact) to 4 (maximum impact). Total scores ranged from 8 (no impact) to 32 (maximum impact).
Time Frame: Baseline, Week 28
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Aripiprazole | Paliperidone
Number analyzed (Participants) | 136 | 132
units on a scale | -1.75 (0.30) | -1.05 (0.32)
Statistical Analysis 1: Comparison: Aripiprazole vs Paliperidone; Test type: Superiority or Other; p = 0.095, Mixed Models Analysis — All secondary endpoints were tested without any hierarchical testing strategy and no adjustment for multiplicity; The model uses an unstructured variance/covariance matrix; Least Squares Mean Difference = -0.695, 95% CI 2-sided [-1.511 to 0.121]

ADVERSE EVENTS:
Time Frame: First dose to end of study (32 weeks)
Groups:
- ARIPIPRAZOLE; PALIPERIDONE: Safety data is based on all patients who received study medicine.
Arm/Group | ARIPIPRAZOLE | PALIPERIDONE
Serious Adverse Events (participants affected / at risk) | 12/144 | 10/137
Other Adverse Events (participants affected / at risk) | 64/144 | 74/137
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ARIPIPRAZOLE (N=144) | PALIPERIDONE (N=137)
Cirrhosis alcoholic (Hepatobiliary disorders) | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Intentional overdose (Injury, poisoning and procedural complications) | 1 | 0
Nasopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Psychotic disorder (Psychiatric disorders) | 5 | 4
Schizophrenia (Psychiatric disorders) | 5 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Suividal ideation (Psychiatric disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ARIPIPRAZOLE (N=144) | PALIPERIDONE (N=137)
Nausea (Gastrointestinal disorders) | 3 | 8
Fatigue (General disorders) | 4 | 7
Injection site pain (General disorders) | 4 | 11
Nasopharyngitis (Infections and infestations) | 6 | 8
Accidental overdose (Injury, poisoning and procedural complications) | 30 | 13 — these events occurred during the oral treatment phase of the study
Weight increased (Investigations) | 13 | 19
Akathisia (Nervous system disorders) | 8 | 6
Dizziness (Nervous system disorders) | 5 | 12
Headache (Nervous system disorders) | 3 | 11
Somnolence (Nervous system disorders) | 9 | 8
Anxiety (Psychiatric disorders) | 8 | 12
Insomnia (Psychiatric disorders) | 17 | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No